CLINICAL TRIAL: NCT00156559
Title: MMR and Varicella Vaccine Responses in Extremely Premature Infants
Brief Title: MMR and Varicella Vaccine in Premature Infants
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Carl D'Angio, Professor, University of Rochester
Other Study IDs: DMID 03-140; N01-AI-25460
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Chickenpox; Rubella; Rubeola; Mumps
Keywords: immunization; vaccine; low birth weight infant; premature infant
MeSH Terms: conditions — Chickenpox; Rubella; Measles; Mumps; Premature Birth

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This research is designed to address the question, "Does the relative deficit in vaccine immunogenicity in extremely premature infants persist beyond the first 6 months of life?" We propose to measure the immunogenicity of varicella and mumps-measles-rubella vaccines in relatively healthy, 12-to-15 month-old children born at <29 weeks gestation, when compared to full-term infants, as measured by the relevant viral serologies.

DETAILED DESCRIPTION:
Title: MMR and Varicella Vaccine Responses in Extremely Premature Infants

Phase: IV

Population: 16 generally healthy premature infants born at < 29 weeks' gestation, < 16 months old from the Rochester area 16 generally healthy full-term infants born at >/= 37 weeks' gestation, < 16 months old from the Rochester area

Number of Sites: University of Rochester

Study Duration: 1.5 - 8.5 months

Description of Agent or Intervention:

Subjects will make 2 study visits. The first, at 15 months of age, will coincide with a routine well child visit. Subjects will have 2 mL of blood drawn at the time of their routine, 15-month MMR, varicella, and pneumococcal conjugate immunizations. At a second study visit 4-6 weeks later, another 2 mL of blood will be drawn.

Objectives:

Primary: We propose to measure the immunogenicity of routinely administered varicella and mumps-measles-rubella vaccines in relatively healthy, 12-to-15 month-old children born at <29 weeks gestation (premature), when compared to that in full-term infants.

Measles titers will be measured by neutralization assay. Mumps and rubella titers will be measured by enzyme-linked florescent immunoassay. Varicella titers will be measured by enzyme linked immunosorbent assay.

Safety will be assessed by parental recall of vaccine-related adverse events and by active, prospective collection of blood-draw-associated adverse events.

Schematic of Study Design:

Subjects will be approached at 9-12 months of age for inclusion, and will consent at this time or at Visit 1

Visit 1 (15 mos):

Preterm N = 16, Full term N = 16, 2 ml blood draw

Routine MMR, varicella vaccines administered by primary pediatrician per standard of care (at Visit 1)

Visit 2 (16 mos):

Preterm N = 16, Full term N = 16, 2 ml blood draw

Varicella, mumps, measles and rubella vaccine titers measured by ELISA

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the inclusion criteria to participate in this study.

1. Premature infant < 29 weeks' gestation at birth or term infant >/= 37 weeks' gestation at birth.
2. Postnatal age < 16 months, 0 days.
3. Has not yet received MMR or varicella vaccines. (There are no restrictions on the administration of other vaccines at the time of MMR/varicella vaccination.)
4. Parental permission.
5. Agreement of primary care pediatrician/ health care provider.
6. Receives primary pediatric care within an approximate 25-mile radius of the University of Rochester.
7. Healthy status at enrollment.

Exclusion Criteria:

1. Known immunodeficiency.
2. Systemic corticosteroid therapy at the time of MMR/varicella vaccination.
3. Requiring oxygen therapy.
4. Clinically significant findings on review of medical history and physical exam determined by the investigator or sub-investigator to be sufficient for exclusion.
5. Any condition determined by the investigator that would interfere with the evaluation of the vaccine or be a potential health risk to the subject.

Ages: 12 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32
Dates: Start 2004-01; Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl T. D'Angio, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Result] D'Angio CT, Boohene PA, Mowrer A, Audet S, Menegus MA, Schmid DS, Beeler JA. Measles-mumps-rubella and varicella vaccine responses in extremely preterm infants. Pediatrics. 2007 Mar;119(3):e574-9. doi: 10.1542/peds.2006-2241. PMID 17332177